CLINICAL TRIAL: NCT02189863
Title: Driving Simulator Study Comparing Two Modes of Presbyopic Correction With Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: M-14-009
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-01

CONDITIONS: Presbyopia
Keywords: Driving Simulator; Air Optix Aqua; AOAMF
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AOAMV, then AOAMF (Other): Lotrafilcon B MV contact lenses worn for 2 weeks in Period 1, followed by lotrafilcon B MF contact lenses worn for 2 weeks in Period 2
  Interventions: Device: Lotrafilcon B MF; Device: Lotrafilcon B MV; Device: Lotrafilcon B SVD; Device: Comfilcon A MF; Device: Habitual contact lenses
- AOAMF, then AOAMV (Other): Lotrafilcon B MF contact lenses worn for 2 weeks in Period 1, followed by lotrafilcon B MV contact lenses worn for 2 weeks in Period 2
  Interventions: Device: Lotrafilcon B MF; Device: Lotrafilcon B MV; Device: Lotrafilcon B SVD; Device: Comfilcon A MF; Device: Habitual contact lenses

INTERVENTIONS:
Device: Lotrafilcon B MF — Multifocal contact lenses worn in both eyes
  Other Names: AIR OPTIX® Aqua Multifocal; AOAMF
Device: Lotrafilcon B MV — Spherical contact lenses worn with 1 eye corrected for distance and 1 eye corrected for near
  Other Names: AIR OPTIX® Aqua; AOAMV
Device: Lotrafilcon B SVD — Spherical contact lenses worn with both eyes corrected for distance
  Other Names: AIR OPTIX® Aqua
Device: Comfilcon A MF — Multifocal contact lenses worn in both eyes
  Other Names: Biofinity® Multifocal
Device: Habitual contact lenses — Contact lenses worn in both eyes per subject's habitual prescription

SUMMARY:
The overall objective of this study is to compare the effect on simulated driving performance of multifocal (MF) versus monovision (MV) soft contact lenses in mid-late presbyopes.

DETAILED DESCRIPTION:
In this crossover study, subjects wore lotrafilcon B MV (AOAMV) and lotrafilcon B MF (AOAMF) soft contact lenses as randomized for 2 weeks each. Subjects were assessed using a standardised driving simulation for each of the two treatments. A fresh pair of lenses was dispensed for the assessment. Subjects also wore lotrafilcon B single vision distance (SVD) and comfilcon A MF contact lenses during Period 1 and Period 2 respectively for an additional same-day assessment. Habitual correction was worn for an acclimatization drive in the driving simulator during Period 1.

ELIGIBILITY:
Inclusion Criteria:

* Current soft contact lens wearers (for 1 month or more) with distance spherical power requirements of +1.00 to + 4.00 diopters (D) or -1.00 to -10.00D, and who have never tried and then failed in monovision or AOAMF.
* Medium to high presbyopia, i.e. spectacle add requirement of +1.50D or more.
* Astigmatism, if present, ≤1.00D in both eyes.
* Distance visual acuity (VA) correctable to 20/30 (+0.2 logMAR) in both eyes.
* Within the normal ranges for binocular vision for distance (8Δ exophoria, ≤8Δ esophoria), vertical phoria = 1.5Δ hypo or hyper.
* Full United Kingdom driving license held for at least 3 years, with at least 2000 miles driven per year.
* Willing to wear study lenses at least 5 days per week.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Existing AIR OPTIX® Multifocal CL user.
* Sphere requirement in the range +0.75 to -0.75D in both eyes.
* Previous refractive surgery.
* Ocular/systemic medical condition or medical treatment contra-indicating contact lens wear or driving simulation.
* Participation in a clinical study within the past 30 days.
* Other protocol-defined exclusion criteria may apply.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Manager, Global Medical Affairs, Vision Care, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 2 investigational sites located in the UK.
Pre-assignment Details: Of the 33 enrolled, 6 participants were exited as screen failures prior to randomization. This reporting group includes all randomized participants who successfully tried at least one study lens (27).
Groups:
- AOAMV, Then AOAMF: Lotrafilcon B MV contact lenses (AOAMV) worn for 2 weeks in Period 1, followed by lotrafilcon B MF contact lenses (AOAMF) worn for 2 weeks in Period 2
Period: First 2 Weeks
Arm/Group | AOAMV, Then AOAMF | AOAMF, Then AOAMV
Started | 12 | 15
Completed | 8 | 13
Not Completed | 4 | 2
Not completed — Motion Sickness | 4 | 2
Period: Second 2 Weeks
Arm/Group | AOAMV, Then AOAMF | AOAMF, Then AOAMV
Started | 8 | 13
Completed | 8 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized participants who successfully tried at least one study lens.
Groups:
- Overall: Lotrafilcon B MV and lotrafilcon B MF contact lenses worn in Period 1 and Period 2, as randomized
Arm/Group | Overall
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Driving Reaction Time to Hazards (as Measured by Time to Brake, in Seconds)
Description: Driving reaction time to hazards was assessed during simulated night time driving and measured as time to brake, in seconds. One eye (study eye) contributed to the analysis. This outcome measure was prespecified for AOAMV and AOAMF.
Time Frame: Week 2, each period
Population: This analysis population includes all randomized subjects in the groups to which they were randomly assigned who successfully completed both study lens follow-up evaluations without a protocol deviation that was documented as impacting the assessment of the hypotheses (Per-Protocol).
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- AOAMV: Lotrafilcon B spherical contact lenses worn with 1 eye corrected for distance and 1 eye corrected for near for 2 weeks
- AOAMF: Lotrafilcon B multifocal contact lenses worn in both eyes for 2 weeks
Arm/Group | AOAMV | AOAMF
Number analyzed (Participants) | 21 | 21
seconds | 1.89 (0.22) | 1.88 (0.19)

2. Secondary Outcome: Standard Deviation of Lateral Positioning
Description: The standard deviation of lateral positioning (staying in the lane) was assessed during simulated night time driving and measured as the distance of deviation from the reference point, in meters. This outcome measure is prespecified for AOAMV and AOAMF.
Time Frame: Week 2, each period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | AOAMV | AOAMF
Number analyzed (Participants) | 21 | 21
meters | 0.35 (0.06) | 0.35 (0.05)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of a subject's participation in the study (up to 4 weeks). This analysis group includes all randomized subjects who successfully tried at least one study lens, based on treatment-specific exposure.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the medical device. Ocular adverse events are presented for both study eye and non-study eye.
Groups:
- Lotra B SVD: Lotrafilcon B spherical contact lenses worn with both eyes corrected for distance during Period 1 for a same-day assessment
- Biofinity MF: Comfilcon A multifocal contact lenses worn in both eyes during Period 2 for a same-day assessment
- Habitual: Contact lenses worn in both eyes per subject's habitual prescription on Day 1, Period 1, for a same-day assessment
Arm/Group | AOAMV | AOAMF | Lotra B SVD | Biofinity MF | Habitual
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23 | 0/23 | 0/21 | 0/27
Other Adverse Events (participants affected / at risk) | 1/25 | 1/23 | 2/23 | 0/21 | 2/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AOAMV (N=25) | AOAMF (N=23) | Lotra B SVD (N=23) | Biofinity MF (N=21) | Habitual (N=27)
Motion sickness (General disorders) | 1 | 1 | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.